CLINICAL TRIAL: NCT01570530
Title: Atorvastatin Using as a Possible Prophylaxis of Postoperative Atrial Fibrillation After Cardiac Surgery
Acronym: PROFACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: End of finantial support
Sponsor: Fundación General Universidad de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROFACE
Record Dates: First submitted 2012-03-01; First posted 2012-04-04 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): Patients treated with atorvastatin
  Interventions: Procedure: Cardiac surgery
- Without Atorvastatin (Other): Patients treated without atorvastatin
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Atorvastatin therapy as prophylaxis against postoperative atrial fibrillation after cardiac surgery
  Arms: Atorvastatin
Procedure: Cardiac surgery — Without atorvastatin therapy as prophylaxis against postoperative atrial fibrillation after cardiac surgery
  Arms: Without Atorvastatin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of atorvastatin therapy (both during preoperative and postoperative period), as prophylaxis against postoperative atrial fibrillation after cardiac surgery, in a valve disease patient population (with or without associated coronary artery disease), with no previous history of atrial fibrillation and not receiving beta-blocking drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 year-old.
2. In sinus rhythm.
3. Affected by valve disease, isolated or associated with coronary artery disease, satisfying requirements for heart surgery under extracorporeal circulation.
4. Women of childbearing potential must use effective contraception and they must commit to maintain it throughout the study.

Exclusion Criteria:

1. Urgent surgery.
2. Surgery due to endocarditis.
3. Patients with previous episodes of atrial fibrillation, although they are in sinus rhythm at hospital admission.
4. Treatment with beta-blockers at time of randomization
5. Severe left ventricular dysfunction with ventricular ejection fraction under 30%.
6. Chronic using of NSAIDs and / or corticosteroids at time of randomization
7. Uncontrolled thyroid disease.
8. Active liver disease and / or history of previous chronic liver disease.
9. Alcoholism.
10. Predisposing factors to statins adverse effects:

    * Increased transaminase levels at baseline (x3 normal value).
    * Renal failure (creatinine levels over 2 mg/dl).
    * Previous diagnosis of myopathy of any etiology.
11. Known hypersensitivity to calcium atorvastatin and / or lactose monohydrate
12. In women of childbearing age, positive pregnancy test the day of inclusion in the study.
13. Not signed informed consent.
14. Inability to understand objectives of the study.

Exclusion criteria of the study once started:

* Withdrawal of patient's consent.
* Modification in liver laboratory parameters (transaminases above three times normal value) and / or creatine-fosfokinase level suggesting adverse effects of statins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative atrial fibrillation(atorvastatin and control groups) | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
  To evaluate the effectiveness of atorvastatin therapy (both during preoperative and postoperative period), as prophylaxis against postoperative atrial fibrillation after cardiac surgery, in a valve disease patient population (with or without associated coronary artery disease), with no previous history of atrial fibrillation and not receiving beta-blocking drugs or statins.

SECONDARY OUTCOMES:
Changes in inflammatory markers values during extracorporeal circulation, and postoperative atrial fibrillation. | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Changes in biochemical markers in both groups. | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Changes in echocardiographic parameters in both groups. | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Frequency, duration, characteristics and risk factors for postoperative atrial fibrillation in patients with valve disease (without history of previous arrhythmia) undergoing cardiac surgery. | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Clinical and hemodynamic consequences of postoperative atrial fibrillation after cardiac surgery. | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Prolongation of in-hospital and Intensive Care Unit (ICU) stay and the need for new drug or interventionism therapies, directly related to its appearance. | Participants will be followed for the duration of hospital day, an expected average of 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Carrascal Hinojal, M.D, Principal Investigator — Hospital Clínico Universitario de Valladolid
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid, Spain